CLINICAL TRIAL: NCT06718062
Title: Non-Inferiority Study of Aliskiren vs Losartan in the Treatment of Hypertension With Hyperuricemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hansung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20241128-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hypertension,Essential; Hyperuricemia
Keywords: Hypertension; Hyperuricemia; Non-inferiority
MeSH Terms: conditions — Essential Hypertension; Hyperuricemia; Hypertension | interventions — aliskiren; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aliskiren Group (Placebo Comparator): Participants in this group will receive Aliskiren (240 mg daily) for the treatment of hypertension combined with hyperuricemia. The medication will be provided by Shenzhen Xinlitai Pharmaceutical Co., Ltd., with the approval number National Drug Approval No. H20138002. The patients will take Aliskiren orally once a day for 3 months. The primary objective is to assess the non-inferiority of Aliskiren in lowering serum uric acid levels, as well as its effects on blood pressure and kidney function.
  Interventions: Drug: Aliskiren
- Losartan Group (Active Comparator): Participants in this group will receive Losartan (100 mg daily) for the treatment of hypertension combined with hyperuricemia. The medication will be provided by Zhejiang Huahai Pharmaceutical Co., Ltd., with the approval number National Drug Approval No. H20143030. The patients will take Losartan orally once a day for 3 months. The goal is to compare the efficacy of Losartan in reducing serum uric acid levels with Aliskiren and evaluate its impact on blood pressure and kidney function.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Aliskiren — Participants in this group will receive Aliskiren (240 mg daily) for the treatment of hypertension combined with hyperuricemia. The medication will be administered orally once a day for 3 months. The drug will be provided by Shenzhen Xinlitai Pharmaceutical Co., Ltd., with the National Drug Approval No. H20138002. The primary objective is to evaluate the non-inferiority of Aliskiren in lowering serum uric acid levels, and its effects on blood pressure and kidney function.
  Arms: Aliskiren Group
Drug: Losartan — Participants in this group will receive Losartan (100 mg daily) for the treatment of hypertension combined with hyperuricemia. The medication will be administered orally once a day for 3 months. The drug will be provided by Zhejiang Huahai Pharmaceutical Co., Ltd., with the National Drug Approval No. H20143030. The goal is to compare the efficacy of Losartan in reducing serum uric acid levels with Aliskiren and evaluate its impact on blood pressure and kidney function.
  Arms: Losartan Group

SUMMARY:
This clinical trial aims to evaluate the non-inferiority of Aliskiren compared to Losartan in the treatment of hypertension combined with hyperuricemia. Hypertension and hyperuricemia often coexist and may exacerbate each other, increasing the risk of cardiovascular and renal complications. Both Aliskiren and Losartan are widely used for managing hypertension, but their effects on serum uric acid levels and renal function are not well understood in this patient population.

This study will involve 66 participants, randomly assigned to receive either Aliskiren (240 mg daily) or Losartan (100 mg daily) for a treatment period of 3 months. The primary outcome will be the change in serum uric acid levels before and after treatment. Secondary outcomes include changes in blood pressure, kidney function (measured by creatinine levels, eGFR), and adverse events.

The primary objective is to demonstrate that Aliskiren is non-inferior to Losartan in lowering serum uric acid levels. Additionally, the study will assess whether Aliskiren, while effectively managing blood pressure, has a lesser impact on kidney function compared to Losartan.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Hypertension
2. Diagnosed with Hyperuricemia
3. Serum uric acid levels between 420 μmol/L and 700 μmol/L
4. Age between 18 and 80 years
5. Able to provide informed consent
6. No history of gout
7. No serious comorbidities such as severe kidney, liver, or cardiovascular diseases

Exclusion Criteria:

1. Diagnosis of Gout
2. History of secondary hypertension
3. Severe organ dysfunction, including liver, kidney, or heart failure
4. History of malignant tumors
5. Severe cognitive disorders or mental illness
6. Pregnant or breastfeeding women
7. Allergy to study medications (Aliskiren or Losartan)
8. Participation in other clinical trials during the study period

Ages: 37 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Uric Acid Levels | Baseline (before treatment) and 3 months
  The primary outcome measure is the change in serum uric acid levels from baseline to the end of treatment (3 months) in both the Aliskiren and Losartan treatment groups. Serum uric acid levels will be measured using the uricase method from 5 mL fasting venous blood samples before and after treatment. This measure will assess the non-inferiority of Aliskiren compared to Losartan in lowering serum uric acid levels in patients with hypertension and hyperuricemia.

SECONDARY OUTCOMES:
Change in Blood Pressure | Baseline (before treatment) and 3 months
  The secondary outcome measure is the change in blood pressure (systolic and diastolic) from baseline to the end of treatment (3 months). Blood pressure will be measured using a sphygmomanometer after the participant has rested for at least 5 minutes, with three measurements taken at 1-minute intervals and the average value used.
Change in Kidney Function | Baseline (before treatment) and 3 months
  Change in Kidney Function The secondary outcome measure is the change in kidney function, creatinine (Cr) ， from baseline to the end of treatment (3 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Chancheng District People's Hospital, Foshan City, Foshan, Guangdong, China